CLINICAL TRIAL: NCT01677026
Title: Data Collection on the ATI Neurostimulation System: SPG Stimulation for Cluster Headache
Status: Completed | Type: Observational
Sponsor: Autonomic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-004
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objectives of the Registry are to:

1. Monitor the transfer of the ATI Neurostimulation System and its safety/clinical performance to a larger number of centers in the post market phase and
2. Collect additional evidence to support reimbursement and clinical acceptance and long term follow up

ELIGIBILITY:
Inclusion Criteria:

* Subject meets CE marked labeling for cluster headache.
* Subject's typical cluster headache bouts last a minimum of 16 weeks, in the opinion of the Investigator.
* Subject agrees to maintain current preventive headache medication regimens (no change in type, frequency or dose except to manage tolerability) from Study Enrollment through the completion of the Therapy Evaluation Period.
* Subject has the ability to read, comprehend and to reliably record information as required by the Protocol.
* Subject is able to provide written informed consent prior to participation in the study.

Exclusion Criteria:

* Subject has had a change in type, dosage or frequency of taking preventive headache medications < one (1) month prior to Study Enrollment.
* Per the CE marked labeling: In the opinion of the Investigator, subject has bony facial deformities, inappropriate surgical anatomy or has had facial surgery in the surgical area on the same side as the planned surgery that would prevent the proper placement of the ATI Neurostimulator.
* Subject has other significant pain problem that might confound the study assessments in the opinion of the Investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who meet the CE marked labeling for cluster headache for the ATI Neurostimulation System.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Character of usability and acceptance of the ATI Neurostimulation System, as evaluated by the following: | Through study completion
  1. Implantation of ATI Neurostimulator within the pterygopalatine fossa
  2. Explant and lead-revision rates and reasons
Characterization of patient response to therapy, as evaluated by the following: | Through study completion
  1. Patient acceptance of the therapy
  2. Responder Analysis, where a responder is any patient who achieves Effective Therapy in at least 50% of evaluable attacks, a 50% attack frequency attack decrease relative to Baseline, or both
  3. Disability and Quality of Life as characterized by the HIT-6 and SF-36v2 compared to Baseline
  4. Subject Overall Evaluation of Therapy
  5. Change in use of acute medications compared to Baseline
  6. Change in preventive medication use and work status compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Arne May, MD, PhD, Principal Investigator — Institut fur systemische Neurowissenschaften, Universitastsklinikum Hamburg-Eppendorf (UKE)
Locations (11):
- Danish Headache Center, Glostrup Municipality, Denmark
- Germany (10):
  - Berlin Charite Hospital, Berlin
  - Neurologische Klinik und Poliklinik, Bochum
  - Headache Center, Dept. Of Neurology, Univ. Duisburg-Essen, Essen
  - Institut fur systemische Neurowissenschaften, Universitastsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Universitatsklinikum Jena Klinik f. Neurologie, Jena
  - Klinik fur Mund-, Kiefer-und Gesichtschirurgie, Rotes, Kassel
  - Migraine- und Kopfschmerzklinik Konigstein, Königstein
  - Neurologie & Kopfschmerzzentrum Munchner Freiheit, Munich
  - University of Munich-Klinikum der Universitat Munchen Neurologische Klinik und Poliklinik, Munich
  - Universitatsklinikum Munster, Klinik und Poliklinik fur Neurologie, Münster